CLINICAL TRIAL: NCT04280367
Title: Childhood Learning and Executive Function Disorders and Risk of Psychosis in the Adulthood
Brief Title: Learning and Executive Function Disorders in Children and Psychosis Risk at Adult-age
Acronym: DYS FUTURS UHR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191093; 2019-A02663-54 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia; Learning Disorders; Executive Function Disorders
Keywords: learning disorders; executive function disorders; psychosis; children; adult-age
MeSH Terms: conditions — Schizophrenia; Learning Disabilities; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Comparator group: Specific learning disorders group
  Interventions: Diagnostic Test: Standardised semi-structured talk; Diagnostic Test: Autistic spectre disorder screening; Diagnostic Test: Anxiety measuring
- neuro-developmental complexed group: Group of neuro-developmental complexe of learning
  Interventions: Diagnostic Test: Standardised semi-structured talk; Diagnostic Test: Autistic spectre disorder screening; Diagnostic Test: Anxiety measuring
- Complexed with anxiety: Disorders in learning with anxiety
  Interventions: Diagnostic Test: Standardised semi-structured talk; Diagnostic Test: Autistic spectre disorder screening; Diagnostic Test: Anxiety measuring

INTERVENTIONS:
Diagnostic Test: Standardised semi-structured talk — Comprehensive assessment of at-risk mental states (CAARMS) will be used.
Diagnostic Test: Autistic spectre disorder screening — Autism-spectrum quotient (AQ) auto-questionnaire will be used.
Diagnostic Test: Anxiety measuring — An inventory for measuring clinical anxiety: Beck Anxiety Inventory (BAI); Liebowitz Social Anxiety Scale.

SUMMARY:
The primary objective of the study aims to study transition toward schizophrenia in patients with learning disorders, and to compare the risk between patients with specific learning disorders, and patients with complexed learning disorders (by two types: patients with other neuro-developmental disorders including executive function disorders, and patients with anxiety).

DETAILED DESCRIPTION:
As secondary objectives, the study aims to:

* argue the clinical predicted markers (neuropsychological) transition toward psychosis.
* test the feasibility and the acceptability of a early diagnosis for a potential applicable guidance for different referent centers of learning in French territory.
* have a better classification of patients with learning disorders in order to target a prospective primary prevention of risk of psychosis via the questionnaires (AQ of Baron-Cohen: Autism-spectrum quotient auto-questionnaire; Inventory of Beck Anxiety Inventory, auto-questionnaire for panic disorder and general anxiety; Liebowitz Social Anxiety Scale).
* improve identification of the early signs and the early emerging psychological diseases intervention management (schizophrenia).
* Psychic disability: prevent and reduce non-seeking care and accompaniment situations, and risk of rupture of care.
* permitting better care of psychosocial rehabilitation with cognitive evaluation.

This study will be conducted in Centre de référence des troubles du langage et des apprentissages, Hôpital Raymond Poincaré, APHP, in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients born between 1990 and 2005, have been cared by Dr Schlumberger in 2014 in the center of language and learning disorders at Raymond Poincaré hospital;
* With severe learning disorders: deficiency in school work, need at least one medical appointment and long-term rehabilitation in the center of language and learning disorders at Raymond Poincaré hospital;
* Affiliated to a social protection schema;
* Written informed consent signed.

Exclusion Criteria:

* Absence of learning disorder;
* Intellectual deficiency;
* Epilepsia;
* Patients who will performed follow-up at Chartres city;
* Patients under guardianship or curatorship;
* Foreign patients under AME schema, a medical help from the state in France.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between 15 and 30 years, suffering learning disorders complicated with two orders: with other neuro-developmental, or with anxiety (vs specific: comparator group).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview | At baseline
  Assessement with Comprehensive Assessment of At-Risk Mental States (CAARMS) during 6 to 90 minutes at the center of Raymond Poincaré hospital.
  The unique collection during the interview, quotation of each patient will be given from the assessement.
  There will be 4 groups by the results: CAARMS negative subjects, vulnerable subjects, attenuated psychosis subjects and subjects with brief and limited intermittent psychotic syndrome. The further statistic comparison will be done between the 3 last groups classified with results of CAARMS.

SECONDARY OUTCOMES:
Autistic screening | At baseline
  Autism-spectrum quotient (AQ) auto-questionnaire will be used to evaluate difficulty in social interaction.
Anxiety measuring | At baseline
  An inventory for measuring clinical anxiety: Beck Anxiety Inventory
Social interaction difficulty evaluation | At baseline
  Liebowitz Social Anxiety Scale as questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emilie SCHLUMBERGER, MD, Principal Investigator — Centre de référence des troubles du langage et des apprentissages, Hôpital Raymond Poincaré, APHP; Albane Mansoux, Study Director — Centre de référence des troubles du langage et des apprentissages, Hôpital Raymond Poincaré, APHP
Locations (1):
- Centre de référence des troubles du langage et des apprentissages, Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No